CLINICAL TRIAL: NCT06460233
Title: Dynamics of Blood Pressure Changes After Bariatric Surgery, Assessed With 24-h Blood Pressure Monitoring
Brief Title: Blood Pressure Changes After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Grzegorz Styczyński, Clinical Professor, Medical University of Warsaw
Other Study IDs: KB/173/2020
Record Dates: First submitted 2024-05-24; First posted 2024-06-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Blood Pressure; Obesity; Bariatric Surgery; Hypertension
Keywords: Hypertension; Obesity; Bariatric surgery
MeSH Terms: conditions — Obesity; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen peripheral blood serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with class III obesity (BMI ≥ 40) or class II obesity (BMI 35-40) with comorbidities: Consecutive patients with class III obesity (BMI ≥ 40kg/m2) or class II obesity (BMI 35-40kg/m2) with comorbidities admitted for bariatric surgery (sleeve gastrectomy)
  Interventions: Procedure: Bariatric surgery - sleeve gastrectomy

INTERVENTIONS:
Procedure: Bariatric surgery - sleeve gastrectomy — Laparoscopic sleeve gastrectomy performed according to the current surgical standards

SUMMARY:
The aim of the study is to assess changes in blood pressure, cardiac function and selected laboratory measurements after bariatric surgery and to find most important factors associated with blood pressure reduction after weight loss.

Description of the study

Patients: consecutive patients with class III obesity (BMI ≥ 40kg/m2) or class II obesity (BMI 35-40kg/m2) with comorbidities, admitted for sleeve gastrectomy

Methods: bedside and 24-hour blood pressure measurement, cardiac ultrasound and laboratory tests performed before surgery and at 1 week, 4 weeks, 6 months and 12 months after bariatric surgery

DETAILED DESCRIPTION:
Pathogenesis of blood pressure reduction associated with weight loss is not established. We hypothesize that monitoring of blood pressure changes after weight loss, with concomitant evaluation of cardiac output and selected biochemical parameters related to blood pressure regulation may help in the understanding of weight loss-associated decrease in blood pressure.

The study protocol include measurement of blood pressure (bedside and 24h blood pressure monitoring), assessment of the cardiac function and biochemistry 1-2 days before laparoscopic sleeve gastrectomy and at the time of routine surgical follow-up visits after surgery ie. one week, one month, six and twelve months. Blood pressure measurements will be performed using automatic oscillometric monitors (OnTrak , Spacelabs,USA). Cardiac evaluation will include an echocardiographic assessment of the systolic and diastolic left ventricular function as well as cardiac output measurement using Doppler method. Biochemistry measures, in addition to routine blood tests needed for surgical follow-up, will include fasting insulin, high sensivity C-reactive protein, cystatin C, and NT-proBNP.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥40kg/m2 or ≥35 kg/m2 with comorbidities

Exclusion Criteria:

* Lack of informed consent
* Expected lack of compliance
* Psychiatric illness
* Previous bariatric surgery
* Severe gastroesophageal reflux disease
* Active neoplastic disease
* Pregnancy
* Chronic atrial fibrillation or other persistent arrhythmia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes all consecutive patients with class III obesity or class II obesity with comorbidities, admitted for bariatric surgery (sleeve gastrectomy) to the Departement of General, Transplant and Liver Surgery, Medical University of Warsaw
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the 24-hour blood pressure at one week after bariatric surgery (sleeve gastrectomy) | 1-2 days before and 7 to 10 days after surgery
  Mean systolic and diastolic blood pressure in mmHg, measured using 24 hour ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Change from baseline in the 24-hour blood pressure at one month after bariatric surgery (sleeve gastrectomy) | 1-2 days before and 28 to 31 days after surgery
  Mean systolic and diastolic blood pressure in mmHg, measured using 24 hour ambulatory blood pressure monitor
Change from baseline in the 24-hour blood pressure at six months after bariatric surgery (sleeve gastrectomy) | 1-2 days before and 5 to 7 months after surgery
  Mean systolic and diastolic blood pressure in mmHg, measured using 24 hour ambulatory blood pressure monitor
Change from baseline in the 24-hour blood pressure at one year after bariatric surgery (sleeve gastrectomy) | 1-2 days before and 11 to 13 months after surgery
  Mean systolic and diastolic blood pressure in mmHg measured using 24 hour ambulatory blood pressure monitor
Change from baseline in bedside blood pressure at one week after bariatric surgery | 1-2 days before and 7 to 10 days after surgery
  Systolic and diastolic blood pressure in mmHg, averaged from two measurements using automatic blood pressure monitor, performed in supine position at the end of echocardiographic study
Change from baseline in bedside blood pressure at one month after bariatric surgery | 1-2 days before and 28 to 31 days after surgery
  Systolic and diastolic blood pressure in mmHg, averaged from two measurements using automatic blood pressure monitor, performed in supine position at the end of echocardiographic study
Change from baseline in bedside blood pressure at six months after bariatric surgery | 1-2 days before and 5 to 7 months after surgery
  Systolic and diastolic blood pressure in mmHg, averaged from two measurements using automatic blood pressure monitor, performed in supine position at the end of echocardiographic study
Change from baseline in bedside blood pressure at one year after bariatric surgery | 1-2 days before and 11 to 13 months after surgery
  Systolic and diastolic blood pressure in mmHg, averaged from two measurements using automatic blood pressure monitor, performed in supine position at the end of echocardiographic study
Change from baseline in cardiac output at one week after bariatric surgery | 1-2 days before and 7 to 10 days after surgery
  Echocardiographic measurement of cardiac output in liters per minute using Doppler method
Change from baseline in cardiac output at one month after bariatric surgery | 1-2 days before and 28 to 31 days after surgery
  Echocardiographic measurement of cardiac output in liters per minute using Doppler method
Change from baseline in cardiac output at six months after bariatric surgery | 1-2 days before and 5 to 7 months after surgery
  Echocardiographic measurement of cardiac output in liters per minute using Doppler method
Change from baseline in cardiac output at one year after bariatric surgery | 1-2 days before and 11 to 13 months after surgery
  Echocardiographic measurement of cardiac output in liters per minute using Doppler method
Change from baseline in the left ventricular systolic function at one week after bariatric surgery | 1-2 days before and 7 to 10 days after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak systolic velocities in meters per second, using tissue Doppler method
Change from baseline in the left ventricular systolic function at one month after bariatric surgery | 1-2 days before and 28 to 31 days after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak systolic velocities in meters per second, using tissue Doppler method
Change from baseline in the left ventricular systolic function at six months after bariatric surgery | 1-2 days before and 5 to 7 months after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak systolic velocities in meters per second, using tissue Doppler method
Change from baseline in the left ventricular systolic function at one year after bariatric surgery | 1-2 days before and 11 to 13 months after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak systolic velocities in meters per second, using tissue Doppler method
Change from baseline in the left ventricular diastolic function at one week after bariatric surgery | 1-2 days before and 7 to 10 days after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak early diastolic velocities in meters per second, using tissue Doppler method, and of the early and late mitral inflow peak velocities in meters per second, using pulse wave Doppler method
Change from baseline in the left ventricular diastolic function at one month after bariatric surgery | 1-2 days before and 28 to 31 days after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak early diastolic velocities in meters per second, using tissue Doppler method, and of the early and late mitral inflow peak velocities in meters per second, using pulse wave Doppler method
Change from baseline in the left ventricular diastolic function at six months after bariatric surgery | 1-2 days before and 5 to 7 months after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak early diastolic velocities in meters per second, using tissue Doppler method, and of the early and late mitral inflow peak velocities in meters per second, using pulse wave Doppler method
Change from baseline in the left ventricular diastolic function at one year after bariatric surgery | 1-2 days before and 11 to 13 months after bariatric surgery
  Echocardiographic measurement of the lateral and medial mitral annulus peak early diastolic velocities in meters per second, using tissue Doppler method, and of the early and late mitral inflow peak velocities in meters per second, using pulse wave Doppler method
Change from baseline in serum fasting insulin level at one week after bariatric surgery | 1-2 days before and 7 to 10 days after bariatric surgery
  Laboratory measurement of serum fasting insulin level in µIU/ml
Change from baseline in serum fasting insulin level at one month after bariatric surgery | 1-2 days before and 28 to 31 days after bariatric surgery
  Laboratory measurement of serum fasting insulin level in µIU/ml
Change from baseline in serum fasting insulin level at six months after bariatric surgery | 1-2 days before and 5 to 7 months after bariatric surgery
  Laboratory measurement of serum fasting insulin level in µIU/ml
Change from baseline in serum fasting insulin level at one year after bariatric surgery | 1-2 days before and 11 to 13 months after bariatric surgery
  Laboratory measurement of serum fasting insulin level in µIU/ml
Change from baseline in serum high- sensivity C-Reactive Protein level at one week after bariatric surgery | 1-2 days before and 7 to 10 days after bariatric surgery
  Laboratory measurement of serum high- sensivity C-Reactive Protein level in mg/l
Change from baseline in serum high- sensivity C-Reactive Protein level at one month after bariatric surgery | 1-2 days before and 28 to 31 days after bariatric surgery
  Laboratory measurement of serum high- sensivity C-Reactive Protein level in mg/l
Change from baseline in serum high- sensivity C-Reactive Protein level at six months after bariatric surgery | 1-2 days before and 5 to 7 months after bariatric surgery
  Laboratory measurement of serum high- sensivity C-Reactive Protein level in mg/l
Change from baseline in serum high- sensivity C-Reactive Protein level at one year after bariatric surgery | 1-2 days before and 11 to 13 months after bariatric surgery
  Laboratory measurement of serum high- sensivity C-Reactive Protein level in mg/l
Change from baseline in serum Cystatin C level at one week after bariatric surgery | 1-2 days before and 7 to 10 days after bariatric surgery
  Laboratory measurement of serum Cystatin C level in mg/l
Change from baseline in serum Cystatin C level at one month after bariatric surgery | 1-2 days before and 28 to 31 days after bariatric surgery
  Laboratory measurement of serum Cystatin C level in mg/l
Change from baseline in serum Cystatin C level at six months after bariatric surgery | 1-2 days before and 5 to 7 months after bariatric surgery
  Laboratory measurement of serum Cystatin C level in mg/l
Change from baseline in serum Cystatin C level at one year after bariatric surgery | 1-2 days before and 11 to 13 months after bariatric surgery
  Laboratory measurement of serum Cystatin C level in mg/l
Change from baseline in serum NT-proBNP level at one week after bariatric surgery | 1-2 days before and 7 to 10 days after bariatric surgery
  Laboratory measurement of serum NT-proBNP level in pg/ml
Change from baseline in serum NT-proBNP level at one month after bariatric surgery | 1-2 days before and 28 to 31 days after bariatric surgery
  Laboratory measurement of serum NT-proBNP level in pg/ml
Change from baseline in serum NT-proBNP level at six months after bariatric surgery | 1-2 days before and 5 to 7 months after bariatric surgery
  Laboratory measurement of serum NT-proBNP level in pg/ml
Change from baseline in serum NT-proBNP level at one year after bariatric surgery | 1-2 days before and 11 to 13 months after bariatric surgery
  Laboratory measurement of serum NT-proBNP level in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Styczynski, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Central Warsaw Medical University Teaching Hospital, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All anonymized patient's data collected during the study will be shared with other researchers who provide methodologically sound proposal
Time Frame: between 3 months and 5 years after the end of the study
Access Criteria: e-mail contact with the principal investigator: grzegorz.styczynski@wum.edu.pl